CLINICAL TRIAL: NCT04128267
Title: Characterization of Central Pain Syndrome in Survivors of Head and Neck Cancer
Brief Title: Central Pain Syndrome in Survivors of Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment/accrual impacted by COVID and technical issues with equipment
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dianne Lou, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC HN 1982
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Results first posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Response to Pain (Experimental): Brain's response to pain using magnetic resonance imaging (MRI)
  Interventions: Device: IPC-1000; Device: Magnetic resonance imaging; Other: Correlative Studies

INTERVENTIONS:
Device: IPC-1000 — Delivers pressure to thumbnail for five seconds at a time
Device: Magnetic resonance imaging — Scan of brain using Magnetic resonance imaging
Other: Correlative Studies — Administration of questionnaires via computer

SUMMARY:
This is a cross-sectional pilot study of head and neck cancer survivors who have completed multi-modal treatment to assess and characterize the presence of distinct pain syndromes.

DETAILED DESCRIPTION:
Primary objectives:

* To correlate structural and functional MRI signature with one of three pain phenotypes in head and neck cancer survivors: 1) no pain, 2) central pain, and 3) nociceptive pain.
* To correlate the presence of chronic systemic symptoms with pain phenotype

Exploratory objectives:

- DNA, RNA, and plasma will be collected for genomic, transcriptomic, and proteomic studies. Results will be vertically integrated along with the results of clinical studies described within this protocol to identify targets for future correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven head and neck cancer
* Patients without a diagnosis of head and neck cancer (up to 10 patients, see below)

  * We anticipate enrolling a total of 75 patients with a history of head and neck cancer who will complete all questionnaires and MRI scanning. We will also recruit up to 10 patients WITHOUT a diagnosis of head and neck cancer to facilitate optimization of the MRI scanning processes. This will allow us to address logistical issues, such as pressure stimulator setup and timing of each scan to be performed.
* Completed multi-modality therapy a minimum of 6 weeks prior to study entry.
* Willing and able to provide informed consent
* All participants must be at least 21 years of age
* Able to speak English

Exclusion Criteria:

* Patients who are pregnant
* Patients who are unable to lie still
* Patients who are unable tolerate pressure stimulator
* Non-MRI compatible devices such as aneurysm clips, cardiac pacemakers or defibrillators, cochlear implants, hardware, or any other implants
* Iron-based tattoos, pieces of metal (bullet, BB, shrapnel) close to or in an important organ (such as the eye), or other non-MRI compatible metal in the body

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Lou, MD, PhD, Principal Investigator — Vanderbilt Medical Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants at Vanderbilt University Medical Center from November 4, 2019 to July 21, 2022. The study stopped early due to low accrual and technical issues with equipment.
Period: Overall Study
Arm/Group | Response to Pain
Started | 32
Completed | 17
Not Completed | 15
Not completed — Withdrawal by Subject | 6
Not completed — Death | 2
Not completed — Disease progression | 1
Not completed — Participant had other medical issues | 4
Not completed — Participant failed to respond to multiple attempts to contact | 2

BASELINE CHARACTERISTICS:
Arm/Group | Response to Pain
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Magnetic Resonance Imaging (MRI) to Correlate With One of Three Pain Phenotypes 1) no Pain, 2) Central Pain, 3) Nociceptive Pain
Description: MRI scan of brain to measure response to stimulated pressure to thumbnail
Time Frame: Approximately 8 weeks
Population: Data were not collected due to the technical issues.
Arm/Group | Response to Pain
Number analyzed (Participants) | 0

2. Primary Outcome: Magnetic Resonance Imaging (MRI) to Correlate Presence of Chronic Systemic Symptoms With Pain Phenotype
Description: MRI scan of brain to measure response to stimulated pressure to thumbnail
Time Frame: Approximately 8 weeks
Population: Data were not collected due to the technical issues.
Arm/Group | Response to Pain
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From date of enrollment until 30 days after completing last study intervention, on average of 3 months
Arm/Group | Response to Pain
All-Cause Mortality (participants affected / at risk) | 3/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/67/NCT04128267/Prot_SAP_002.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT04128267/ICF_001.pdf